CLINICAL TRIAL: NCT02687685
Title: Randomized Clinical Trial of Immediate Skin to Skin Contact (SSC) at Birth, Early vs. Immediate, on the Duration of Exclusive Human Lactation in Full-term Newborns Treated at the Universidad de La Sabana Clinic
Brief Title: Clinical Trial of Immediate Skin to Skin Contact at Birth Early vs. Immediate (CPPITLH)
Acronym: CPPITLH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidad de la Sabana (Other)
Responsible Party: Principal Investigator, Oscar Andrés Gamboa Garay, School of Medicine Professor, Universidad de la Sabana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Acta 313 05-09-2015
Record Dates: First submitted 2016-02-02; First posted 2016-02-22 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Breast Feeding
Keywords: Skin to Skin Contact; Infant, Newborn
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skin to skin contact immediate (Experimental): At birth, the baby will be placed and dried on the breast of his mother where thermoregulation manoeuvres will be applied and once the cord clamping procedure has taken place; the baby will be left in SSC with the mother where the immediate neonatal adaptation interventions will take place. Mother and baby will be left in SSC for at least one hour or until the baby has completed its first lactation properly. Once completed, the baby will be taken to the heat lamp to perform and complete all the newborn mediate adaptation interventions. If the mother expresses the desire to continue in SSC, it will be allowed again after these interventions. During immediate SSC, mother and baby receive continuous monitoring by the health staff
  Interventions: Other: Skin to skin contact immediate
- skin to skin contact early (Active Comparator): At birth, the baby will be dried and placed on the abdomen and chest of his mother where thermoregulation manoeuvres are applied once there is an indication that the cord clamp procedure has been completed. At this time the baby will go to the radiant heat lamp in order to complete all newborn adaptation interventions. Once stable, the mother and the baby who has 60 minutes of life, will proceed with the initiation of SSC for at least one hour or until the baby has completed the first lactation adequately; SSC will be allowed to continue if the mother expresses a desire to do so. During SSC the mother and baby will receive monitoring by health personnel
  Interventions: Other: skin to skin contact early

INTERVENTIONS:
Other: Skin to skin contact immediate — Immediate SSC (intervention group) At birth, the baby will be dried and placed at the mother's breast where thermoregulation maneuvers will be applied and, once cord clamping has taken place, the baby will be left in SSC with the mother where the immediate neonatal adaptation interventions will take place. Mother and baby will be left in SSC for at least 1 h or until the baby has completed its first lactation properly. Once completed, the baby will be taken to the heat lamp to perform and complete all the newborn mediate adaptation interventions. If the mother expresses the desire to continue in SSC, this will be allowed again after these interventions. During immediate SSC, mother and baby will receive continuous monitoring by the health staff.
  Arms: Skin to skin contact immediate
Other: skin to skin contact early — Early SSC group (control group) At birth, the baby will be dried and placed on the abdomen and chest of their mother where thermoregulation maneuvers are applied once cord clamping has been completed. At this time, the baby will placed under the radiant heat lamp in order to complete all newborn adaptation interventions. Once stable, the mother and the baby will proceed with the initiation of SSC for at least 1 h or until the baby has completed the first lactation adequately; SSC will be allowed to continue if the mother expresses a desire to do so. During SSC, the mother and baby will receive monitoring by health personnel. All adaptation interventions, mediate and immediate, in the newborn will take place under the radiant heat lamp during the first postnatal hour.
  Arms: skin to skin contact early

SUMMARY:
SUMMARY: Human lactation is a simple, cost-effective strategy contributing to infant and maternal mortality control. Skin to skin contact (SSC), is an immediate postpartum period strategy that has proven to benefit the initiation and continuation of human lactation and decreased hospitalization during the first week of life. This study aims to determine the effect of the initiation of SSC at birth (immediate vs. early) in healthy, full term newborns treated at Universidad de La Sabana Clinic, on the duration of exclusive human lactation.

Research question: What is the effect of immediate SSC at birth (immediate vs. early) on the duration of exclusive human lactation in full-term newborns treated at the Universidad de La Sabana Clinic?

Methodology: A random blind clinical trial was performed in which full-term healthy newborns that are attended at the Universidad de La Sabana Clinic are included. The blind participants will be those persons measuring the results and analysing the data. The sample size is calculated for a type I error of 5%, a two tailed type II error of 20%, therefore estimating percentage losses of 30%; 150 infants were included per group. Randomization will be performed using permuted, size 6 blocks. Descriptive analysis will be conducted using central tendency and dispersion measurements. A bivariate analysis will be performed to determine which variables are associated with exclusive human lactation at 6 months. For continuous variables, the Student t- test will be used for independent samples or the Wilcoxon rank sum test, in case the assumptions of normality for the t-tests are not fulfilled. The assumption of normality will be evaluated with the Shapiro Wilk and Kolmogorov-Smirnov test. Categorical variables in contingency tables will be constructed, assessing independence between variables with the Chi-square test or Fisher's exact test when the assumption of the number of cases is not met by the cells in the contingency tables, times two. It will be calculated as a measurement of the effect of relative risk (RR) with confidence intervals; the adjusted measurements will be calculated using a multivaried regression Poisson model, variables with significant results will be used in the bivariate analysis and those with biological plausibility used for the adjustment. The analysis will be carried out for a two-tailed type I error level of 5%. The Stata 11 program will be used for the data analysis. An interim analysis will be performed upon submission of half of the expected events (106), setting limits for early termination of the trial according to the method proposed by Pampallona and Tsiatis (1994).

Intervention: There will be 2 SSC randomization groups, early vs. immediate. After completing the neonatal adaptation process and according to the group assignment, it will proceed to leave the newborn with the mother in accommodation. Prior to discharge, the IBFAT scale will be applied. Monitoring will initially be performed with a face valuation between 3 and 10 days of life, then monthly telephone calls for 6 months to verify the status of human lactation.

Results: To determine whether early versus immediate SSC has an impact on the duration of exclusive human lactation.

ELIGIBILITY:
Inclusion Criteria:

* Infants of mothers who express before the birth, their desire to breastfeed their newborn baby.
* Infants born between 7:00 am and 5:00 pm Monday through Friday in the USC.
* Full-term newborns defined by obstetric method and confirmed by paediatric method (Ballard), between 37 and 42 weeks of gestation, with appropriate weight for gestational age (between 10th and 90th percentiles for gestational age).
* Vaginal birth.
* Do not require basic or advanced neonatal resuscitation manoeuvres.
* Healthy and stable cardiorespiratory at birth.
* Have been permitted to room with the mother.

Exclusion Criteria:

* Mothers and newborns that present absolute or relative contraindications for human lactation.
* Multiple births and pregnancies.
* Mothers with postpartum complications that limit the onset of human lactation.
* Major congenital malformations that prevent human lactation.

Max Age: 60 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Exclusive human lactation | Through study completion, an average of 6 months
  Exclusive human lactation for 3 or more months. Exclusive human lactation is defined as: the time in months of human lactation as the only food source without having received other liquids or solid foods (except drugs and / or vitamins)

SECONDARY OUTCOMES:
Human lactation capacity in the newborn | within the first 24 hours of life
  Human lactation capacity in the newborn within the first 24 hours of life by IBFAT Scale
Maternal satisfaction with breastfeeding | First 24 hours
  Maternal satisfaction with breastfeeding in the first 24 hours according to the IBFAT Scale
Evolution of birth weight | First week of life
  Evolution of birth weight in the first week of life.
The need for hospitalization in the neonatal care unit | First week of life
  The need for hospitalization in the neonatal care unit in the first week of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de la Samaritana Unidad Funcional Zipaquira, Zipaquirá, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: Yes
the committee required each month informations about adverse events and informs of recruitment each six months

REFERENCES:
- [Derived] Agudelo SI, Molina CF, Gamboa OA, Acuna E. Comparison of the Effects of Different Skin-to-Skin Contact Onset Times on Breastfeeding Behavior. Breastfeed Med. 2021 Dec;16(12):971-977. doi: 10.1089/bfm.2021.0134. Epub 2021 Sep 7. PMID 34494889
- [Derived] Agudelo SI, Gamboa OA, Acuna E, Aguirre L, Bastidas S, Guijarro J, Jaller M, Valderrama M, Padron ML, Gualdron N, Obando E, Rodriguez F, Buitrago L. Randomized clinical trial of the effect of the onset time of skin-to-skin contact at birth, immediate compared to early, on the duration of breastfeeding in full term newborns. Int Breastfeed J. 2021 Apr 13;16(1):33. doi: 10.1186/s13006-021-00379-z. PMID 33849584
- [Derived] Agudelo S, Gamboa O, Rodriguez F, Cala S, Gualdron N, Obando E, Padron ML. The effect of skin-to-skin contact at birth, early versus immediate, on the duration of exclusive human lactancy in full-term newborns treated at the Clinica Universidad de La Sabana: study protocol for a randomized clinical trial. Trials. 2016 Oct 26;17(1):521. doi: 10.1186/s13063-016-1587-7. PMID 27782829